CLINICAL TRIAL: NCT00532779
Title: A Multicenter, Randomized, Double Blind, Placebo Controlled Study Comparing the Safety and Efficacy of Two Doses of Naltrexone Sustained Release (SR)/Bupropion Sustained Release (SR) and Placebo in Obese Subjects
Brief Title: A Study of the Safety and Efficacy of Two Doses of Naltrexone SR/Bupropion SR and Placebo in Overweight and Obese Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Orexigen Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NB-301; COR-I (Other: Orexigen Therapeutics, Inc.)
Record Dates: First submitted 2007-09-19; First posted 2007-09-20 (Estimated); Results first posted 2014-11-21 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Obesity; Overweight
Keywords: Obesity; Antiobesity agents; Antiobesity drugs; Overweight drug therapy; Obese drug therapy; Weight loss drug effects; Bupropion administration and dosage; Naltrexone administration and dosage; Double blind method; Combination drug therapy; Delayed action preparations
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- NB16 (Experimental): Naltrexone SR 16 mg/Bupropion SR 360 mg /day with ancillary therapy
  Interventions: Drug: Naltrexone SR 16 mg/Bupropion SR 360 mg /day; Behavioral: Ancillary therapy
- NB32 (Experimental): Naltrexone SR 32 mg/Bupropion SR 360 mg /day with ancillary therapy
  Interventions: Drug: Naltrexone SR 32 mg/Bupropion SR 360 mg /day; Behavioral: Ancillary therapy
- Placebo (Placebo Comparator): Placebo with ancillary therapy
  Interventions: Drug: Placebo; Behavioral: Ancillary therapy

INTERVENTIONS:
Drug: Naltrexone SR 16 mg/Bupropion SR 360 mg /day
  Other Names: NB16
  Arms: NB16
Drug: Naltrexone SR 32 mg/Bupropion SR 360 mg /day
  Other Names: NB32
  Arms: NB32
Drug: Placebo
  Arms: Placebo
Behavioral: Ancillary therapy — Ancillary therapy consisting of diet instruction, advice on behavior modification, and exercise counseling

SUMMARY:
The purpose of this study is to determine whether 2 doses of the combination of naltrexone SR and bupropion SR are safe and effective in the treatment of obesity.

DETAILED DESCRIPTION:
Two Phase II clinical trials demonstrated that a combination of bupropion SR and naltrexone is associated with greater weight loss than bupropion SR alone, naltrexone alone, or placebo in subjects with uncomplicated obesity. The current study investigated the safety and efficacy of 2 doses of the combination of naltrexone SR and bupropion SR compared to placebo in obese subjects with uncomplicated obesity and in those with overweight/obesity and hypertension and/or dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Female and male subjects, 18 to 65 years of age;
* Have BMI ≥30 and ≤45kg/m² for subjects with uncomplicated obesity, and BMI of ≥27 and ≤45kg/m² for subjects with obesity and controlled hypertension and/or dyslipidemia;
* Normotensive (systolic ≤140 mm Hg; diastolic ≤90 mm Hg). Anti-hypertensive medications are allowed with the exception of alpha-adrenergic blockers and clonidine; medical regimen must be stable for at least 6 weeks prior to randomization;
* Medications for treatment of dyslipidemia are allowed as long as medical regimen has been stable for at least 6 weeks prior to randomization;
* Free of opioid medication for 7 days prior to randomization;
* No clinically significant abnormality of serum albumin, blood urea nitrogen, creatinine, bilirubin, sodium, potassium, chloride, calcium or phosphorus;
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) within 2.5 x upper limit of normal range (ULN);
* No clinically significant abnormality of hematocrit, white blood cell (WBC) count, white cell differential, or platelets;
* Fasting glucose < 126 mg/dL on no hypoglycemic agents, fasting triglycerides <400 mg/dL;
* No clinically significant abnormality on urinalysis;
* TSH within normal limits or normal T3, if TSH is below normal limits;
* Negative serum pregnancy test in women of child-bearing potential;
* Negative urine drug screen;
* IDS-SR scores < 2 on items 5 (sadness), 6 (irritability), 7 (anxiety/tension) and 18 (suicidality), and IDS-SR total score < 30;
* Women of child bearing potential had to be non-lactating and agree to use effective contraception throughout the study period and 30 days after discontinuation of study drug;
* Able to comply with all required study procedures and schedule;
* Able to speak and read English;
* Willing and able to give written informed consent.

Exclusion Criteria:

* Obesity of known endocrine origin (e.g., untreated hypothyroidism, Cushing's syndrome, established Polycystic Ovary Syndrome);
* Serious medical conditions (including but not limited to ongoing renal or hepatic insufficiency, Class III or IV congestive heart failure; myocardial infarction, history of angina pectoris, claudication, or acute limb ischemia within the previous 6 months; lifetime history of stroke);
* History of malignancy within the previous 5 years with exception of non-melanoma skin cancer or surgically cured cervical cancer;
* A lifetime history of serious psychiatric illness, including lifetime history of bipolar disorder, schizophrenia or other psychosis, bulimia, or anorexia nervosa;
* Current serious psychiatric illness including severe personality disorder, (e.g. borderline or antisocial), current severe major depressive disorder, recent (previous 6 months) suicide attempt, current active suicidal ideation, or recent hospitalization due to psychiatric illness;
* A response to bipolar disorder questions indicating the presence of bipolar disorder;
* In need of medications for the treatment of a psychiatric disorder (with the exception of short-term insomnia) within the previous 6 months prior to randomization;
* History of drug or alcohol abuse or dependence (with the exception of nicotine dependence) within 1 year prior to study initiation;
* Type 1 or Type 2 diabetes mellitus;
* Screening ECG with a corrected QT interval by the method of Bazett (QTcB) >450 msec (men) and > 470 millisecond (msec) (women) or the presence of any clinically significant cardiac abnormalities, including but not limited to patterns consistent with myocardial ischemia, electrolyte abnormalities, or atrial or ventricular dysrhythmia or significant conduction abnormalities;
* Excluded concomitant medications: any psychotropic agents (including antipsychotic, antidepressant, anxiolytic, mood stabilizer, anticonvulsant agents or agents for the treatment of Attention Deficit Disorder) with the exception of low dose benzodiazepine or hypnotic agents for the treatment of insomnia (up to 2 mg lorazepam/day or equivalent dose of a benzodiazepine or hypnotic agent); any anorectic or weight loss agents; any over-the-counter dietary supplements or herbs with psychoactive, appetite or weight effects; alpha-adrenergic blockers; dopamine agonists; clonidine; coumadin; theophylline; cimetidine; oral corticosteroids; cholestyramine, cholestypol, Depo Provera®; smoking cessation agents; use of opioid or opioid-like medications, including analgesics and antitussives;
* History of surgical or device (e.g., gastric banding) intervention for obesity;
* History of seizures of any etiology, or of predisposition to seizures (e.g., history of cerebrovascular accident, head trauma with ≥5 minutes loss of consciousness, concussion symptoms lasting ≥15 minutes, brain surgery, skull fracture, subdural hematoma, or febrile seizures);
* History of treatment with bupropion or naltrexone within the preceding 12 months;
* History of hypersensitivity or intolerance to bupropion or naltrexone;
* Initiation or discontinuation of tobacco products including inhaled tobacco (such as cigarettes, cigars, pipes, etc), chewing tobacco or snuff in the 3 months prior to randomization or planned during study participation. Use of nicotine replacement products (nicotine gum, patch) during study participation was not allowed;
* Use of drugs, herbs, or dietary supplements believed to significantly affect body weight or participation in a weight loss management program within one month prior to randomization;
* Loss or gain of more than 4.0 kilograms within 3 months prior to randomization;
* Pregnant or breast-feeding women or planning to become pregnant during the study period or within 30 days of discontinuing study drug;
* Planned surgical procedure that can impact the conduct of the study;
* Use of investigational drug, device or procedure within the previous 30 days;
* Participation in any previous clinical trial sponsored by Orexigen Therapeutics;
* Any condition which in the opinion of the investigator makes the subject unsuitable for inclusion in the study;
* Investigators, study personnel, sponsor representatives and their immediate families.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1742 (Actual)
Dates: Start 2007-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (34):
- United States (34):
  - Radiant Research, Birmingham, Alabama
  - SelfCenter, PC, Fairhope, Alabama
  - Radiant Research, Phoenix Southeast, Chandler, Arizona
  - Advanced Clinical Research Institute, Anaheim, California
  - Advance Clinical Research Institute, Orange, California
  - Scripps Clinic Del Mar, San Diego, California
  - VA San Diego Healthcare System, San Diego, California
  - Miami Research Associates, Miami, Florida
  - University Clinical Research, Pembroke Pines, Florida
  - Georgia Clinical Research, Atlanta, Georgia
  - CSRA Partners in Health, Inc, Augusta, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Radiant Research, Chicago, Illinois
  - Welborn Clinic, Evansville, Indiana
  - Radiant Research Kansas City, Overland Park, Kansas
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Medical Research Institute, Slidell, Louisiana
  - Health Trends Research, LLC, Baltimore, Maryland
  - FutureCare Studies, Springfield, Massachusetts
  - Center for Nutrition and Metabolic Disorders, Reno, Nevada
  - Center for Nutrition and Preventive Medicine, Charlotte, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Central Ohio Nutrition Center, Inc., Columbus, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Summit Research Network (Oregon), Inc., Portland, Oregon
  - Internal Medicine Associates of Cordova, Cordova, Tennessee
  - Jackson Clinic, PA, Jackson, Tennessee
  - Covance Clinical Research Unit Austin, Austin, Texas
  - Radiant Research, Dallas, Texas
  - Baylor Endocrine Center, Dallas, Texas
  - Radiant Research, San Antonio, Texas
  - Oakwell Clinical Research, San Antonio, Texas

REFERENCES:
- [Result] Greenway FL, Fujioka K, Plodkowski RA, Mudaliar S, Guttadauria M, Erickson J, Kim DD, Dunayevich E; COR-I Study Group. Effect of naltrexone plus bupropion on weight loss in overweight and obese adults (COR-I): a multicentre, randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2010 Aug 21;376(9741):595-605. doi: 10.1016/S0140-6736(10)60888-4. Epub 2010 Jul 29. PMID 20673995

RESULTS

PARTICIPANT FLOW:
Groups:
- NB16: Naltrexone SR 16 mg/Bupropion SR 360 mg /day
- NB32: Naltrexone SR 32 mg/Bupropion SR 360 mg /day
- Placebo: Placebo
Period: Overall Study
Arm/Group | NB16 | NB32 | Placebo
Started | 578 | 583 | 581
Completed | 284 | 296 | 290
Not Completed | 294 | 287 | 291
Not completed — Adverse Event | 122 | 112 | 56
Not completed — Lost to Follow-up | 76 | 65 | 66
Not completed — Withdrawal by Subject | 63 | 60 | 90
Not completed — Lack of Efficacy | 12 | 12 | 40
Not completed — Protocol Violation | 5 | 9 | 7
Not completed — Pregnancy | 2 | 5 | 3
Not completed — Death | 0 | 1 | 0
Not completed — Drug noncompliance, moved, other | 14 | 23 | 29

BASELINE CHARACTERISTICS:
Population: All randomized subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | NB16 | NB32 | Placebo | Total
Number analyzed (Participants) | 578 | 583 | 581 | 1742
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.35 (11.25) | 44.41 (11.14) | 43.66 (11.14) | 44.14 (11.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 490 | 496 | 496 | 1482
  Male | 88 | 87 | 85 | 260
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 13 | 18 | 17 | 48
  Asian | 4 | 6 | 4 | 14
  Native Hawaiian or Other Pacific Islander | 6 | 5 | 4 | 15
  Black or African American | 122 | 106 | 110 | 338
  White | 427 | 440 | 440 | 1307
  Other | 6 | 8 | 6 | 20
Weight [Mean (Standard Deviation); unit: kg] | 99.49 (14.76) | 99.70 (15.88) | 99.45 (14.31) | 99.55 (14.99)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 36.22 (4.28) | 36.10 (4.35) | 36.18 (4.00) | 36.17 (4.21)

OUTCOME MEASURES:

1. Primary Outcome: Co-primary: Body Weight- Mean Percent Change
Time Frame: Baseline, 56 weeks
Population: Modified ITT (Full Analysis Set): Included all subjects who were randomized, had a baseline weight measurement, and had at least one post-baseline weight measurement while on study drug. Missing data were imputed with the LOCF method.
Measure: Least Squares Mean (Standard Error); unit: percentage of body weight
Arm/Group | NB16 | NB32 | Placebo
Number analyzed (Participants) | 471 | 471 | 511
percentage of body weight | -5.00 (0.31) | -6.14 (0.31) | -1.33 (0.30)
Statistical Analysis 1: Comparison: NB16 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -3.67, 95% CI [-4.50 to -2.85]
Statistical Analysis 2: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -4.81, 95% CI 2-sided [-5.63 to -3.99]

2. Primary Outcome: Co-primary: Body Weight- Proportion of Subjects With ≥5% Decrease
Time Frame: Baseline, 56 weeks
Population: Modified ITT: Included all subjects who were randomized, had a baseline weight measurement, and had at least one post-baseline weight measurement while on study drug. Missing data were imputed with the LOCF method.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NB16 | NB32 | Placebo
Number analyzed (Participants) | 471 | 471 | 511
percentage of participants | 39.49 [35.08 to 43.91] | 47.98 [43.47 to 52.49] | 16.44 [13.22 to 19.65]
Statistical Analysis 1: Comparison: NB16 vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.42, 95% CI [2.52 to 4.63]
Statistical Analysis 2: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.86, 95% CI [3.60 to 6.57]

3. Secondary Outcome: Body Weight- Proportion of Subjects With ≥10% Decrease
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | NB16 | NB32 | Placebo
Number analyzed (Participants) | 471 | 471 | 511
Percentage of participants | 20.17 [16.55 to 23.79] | 24.63 [20.74 to 28.52] | 7.44 [5.16 to 9.71]
Statistical Analysis 1: Comparison: NB16 vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.21, 95% CI 2-sided [2.14 to 4.81]
Statistical Analysis 2: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.19, 95% CI 2-sided [2.82 to 6.23]

4. Secondary Outcome: Change in Waist Circumference
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | NB16 | NB32 | Placebo
Number analyzed (Participants) | 342 | 356 | 348
cm | -5.04 (0.43) | -6.24 (0.42) | -2.46 (0.43)
Statistical Analysis 1: Comparison: NB16 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -2.58, 95% CI 2-sided [-3.74 to -1.43]
Statistical Analysis 2: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -3.78, 95% CI 2-sided [-4.93 to -2.64]

5. Secondary Outcome: Change in Fasting HDL Cholesterol Levels
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | NB16 | NB32 | Placebo
Number analyzed (Participants) | 333 | 359 | 345
mg/dL | 3.36 (0.47) | 3.42 (0.45) | -0.06 (0.47)
Statistical Analysis 1: Comparison: NB16 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = 3.42, 95% CI 2-sided [2.17 to 4.66]
Statistical Analysis 2: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = 3.48, 95% CI 2-sided [2.26 to 4.70]

6. Secondary Outcome: Change in Fasting Triglycerides Levels, Using Log-transformed Data
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | NB16 | NB32 | Placebo
Number analyzed (Participants) | 333 | 359 | 345
percent change | -7.96 [-11.35 to -4.44] | -12.69 [-15.79 to -9.47] | -3.08 [-6.62 to 0.60]
Statistical Analysis 1: Comparison: NB16 vs Placebo; Test type: Superiority or Other; p = 0.046, ANCOVA; Mean Difference (Net) = -4.88
Statistical Analysis 2: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -9.61

7. Secondary Outcome: Change in IWQOL-Lite Total Scores
Description: IWQOL-Lite= Impact of Weight on Quality of Life-Lite Questionnaire Total score is based on a scale from 0 to 100, with 0 representing the poorest and 100 the best quality of life and where a score of 71-79 indicates moderate impairment
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NB16 | NB32 | Placebo
Number analyzed (Participants) | 422 | 417 | 468
units on a scale | 11.68 (0.54) | 12.69 (0.54) | 8.55 (0.51)
Statistical Analysis 1: Comparison: NB16 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = 3.13, 95% CI 2-sided [1.72 to 4.54]
Statistical Analysis 2: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = 4.14, 95% CI 2-sided [2.73 to 5.56]

8. Secondary Outcome: Change in High-sensitivity C Reactive Protein (Hs-CRP) Levels, Using Log-transformed Data
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | NB16 | NB32 | Placebo
Number analyzed (Participants) | 331 | 353 | 340
percent change | -28.02 [-34.09 to -21.39] | -28.98 [-34.79 to -22.65] | -16.66 [-23.68 to -9.00]
Statistical Analysis 1: Comparison: NB16 vs Placebo; Test type: Superiority or Other; p = 0.016, ANCOVA; Mean Difference (Net) = -11.36
Statistical Analysis 2: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p = 0.008, ANCOVA; Mean Difference (Net) = -12.32

9. Secondary Outcome: Change in Fasting Insulin Levels, Using Log-transformed Data
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | NB16 | NB32 | Placebo
Number analyzed (Participants) | 309 | 344 | 326
percent change | -11.84 [-17.28 to -6.05] | -17.14 [-21.96 to -12.02] | -4.57 [-10.35 to 1.58]
Statistical Analysis 1: Comparison: NB16 vs Placebo; Test type: Superiority or Other; p = 0.063, ANCOVA; Mean Difference (Net) = -7.27
Statistical Analysis 2: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -12.57

10. Secondary Outcome: Change in Fasting Blood Glucose Levels
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | NB16 | NB32 | Placebo
Number analyzed (Participants) | 336 | 361 | 348
mg/dL | -2.39 (0.57) | -3.24 (0.55) | -1.30 (0.56)
Statistical Analysis 1: Comparison: NB16 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = -1.09, 95% CI 2-sided [-2.60 to 0.42]
Statistical Analysis 2: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p = 0.010, ANCOVA; Mean Difference (Net) = -1.94, 95% CI 2-sided [-3.42 to -0.46]

11. Secondary Outcome: Change in HOMA-IR Levels, Using Log-transformed Data
Description: HOMA-IR= Homeostasis Model Assessment-Insulin Resistance
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | NB16 | NB32 | Placebo
Number analyzed (Participants) | 305 | 341 | 325
percent change | -14.33 [-20.13 to -8.10] | -20.19 [-25.26 to -14.78] | -5.90 [-12.11 to 0.74]
Statistical Analysis 1: Comparison: NB16 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = -8.43
Statistical Analysis 2: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -14.29

12. Secondary Outcome: Change in Question 19 From 21-Item COE (Control of Eating) Questionnaire
Description: Question 19: Generally, how difficult has it been to control your eating? Scoring: 0=not at all difficult; 100=extremely difficult
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NB16 | NB32 | Placebo
Number analyzed (Participants) | 410 | 409 | 453
units on a scale | -12.49 (1.10) | -14.52 (1.09) | -8.68 (1.04)
Statistical Analysis 1: Comparison: NB16 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = -3.81, 95% CI 2-sided [-6.68 to -0.94]
Statistical Analysis 2: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -5.84, 95% CI 2-sided [-8.71 to -2.98]

13. Secondary Outcome: Change in Fasting LDL Cholesterol Levels
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | NB16 | NB32 | Placebo
Number analyzed (Participants) | 332 | 358 | 345
mg/dL | -3.67 (1.21) | -4.41 (1.17) | -3.28 (1.20)
Statistical Analysis 1: Comparison: NB16 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = -0.39, 95% CI 2-sided [-3.62 to 2.84]
Statistical Analysis 2: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p = 0.484, ANCOVA; Mean Difference (Net) = -1.13, 95% CI 2-sided [-4.29 to 2.04]

14. Secondary Outcome: Change in Systolic Blood Pressure
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | NB16 | NB32 | Placebo
Number analyzed (Participants) | 471 | 471 | 511
mm Hg | 0.29 (0.40) | -0.11 (0.41) | -1.94 (0.39)
Statistical Analysis 1: Comparison: NB16 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = 2.23, 95% CI 2-sided [1.16 to 3.30]
Statistical Analysis 2: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = 1.83, 95% CI 2-sided [0.76 to 2.90]

15. Secondary Outcome: Change in Diastolic Blood Pressure
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | NB16 | NB32 | Placebo
Number analyzed (Participants) | 471 | 471 | 511
mm Hg | 0.09 (0.29) | 0.04 (0.29) | -0.86 (0.28)
Statistical Analysis 1: Comparison: NB16 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = 0.96, 95% CI 2-sided [0.19 to 1.73]
Statistical Analysis 2: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = 0.90, 95% CI 2-sided [0.13 to 1.67]

16. Secondary Outcome: Change in IDS-SR Total Scores
Description: IDS-SR= Inventory of Depressive Symptoms-Subject Rated IDS-SR total score is based on 30 items. The total score can range from 0-84, with 0 being no depressive symptoms and 84 being very severe depressive symptoms. A total score ≤ 13 indicates no depression.
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NB16 | NB32 | Placebo
Number analyzed (Participants) | 471 | 470 | 511
units on a scale | 0.02 (0.21) | -0.27 (0.21) | -0.72 (0.20)
Statistical Analysis 1: Comparison: NB16 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = 0.74, 95% CI 2-sided [0.19 to 1.28]
Statistical Analysis 2: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = 0.46, 95% CI 2-sided [-0.09 to 1.00]

17. Secondary Outcome: Change in Food Craving Inventory Sweets Subscale Score
Description: The Food Craving Inventory is a 33-item self-report measure designed to assess specific food cravings and is organized into 4 subscales (high fats, sweets, carbohydrates/starches, and fast-food fats). A craving was defined as an intense desire to consume a particular food (or food type) that was difficult to resist over the past month. Subjects rated their frequency of cravings for each of the 33 items using a 5-point scale, where 1=never, 2=rarely, 3=sometimes, 4=often, and 5=always. The sweets subscale consisted of 8 items and the score ranges from 8 (better outcome) to 40 (worse outcome).
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NB16 | NB32 | Placebo
Number analyzed (Participants) | 423 | 418 | 470
units on a scale | -2.08 (0.21) | -2.62 (0.21) | -2.77 (0.20)
Statistical Analysis 1: Comparison: NB16 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = 0.69, 95% CI 2-sided [0.14 to 1.23]
Statistical Analysis 2: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = 0.15, 95% CI 2-sided [-0.40 to 0.69]

18. Secondary Outcome: Change in Food Craving Inventory Carbohydrates Subscale Score
Description: The Food Craving Inventory is a 33-item self-report measure designed to assess specific food cravings and is organized into 4 subscales (high fats, sweets, carbohydrates/starches, and fast-food fats). A craving was defined as an intense desire to consume a particular food (or food type) that was difficult to resist over the past month. Subjects rated their frequency of cravings for each of the 33 items using a 5-point scale, where 1=never, 2=rarely, 3=sometimes, 4=often, and 5=always. The carbohydrates subscale consisted of 8 items and the score ranges from 8 (better outcome) to 40 (worse outcome).
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NB16 | NB32 | Placebo
Number analyzed (Participants) | 423 | 418 | 469
units on a scale | -1.85 (0.20) | -2.11 (0.20) | -1.84 (0.19)
Statistical Analysis 1: Comparison: NB16 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = -0.00, 95% CI 2-sided [-0.53 to 0.53]
Statistical Analysis 2: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = -0.27, 95% CI 2-sided [-0.80 to 0.27]

ADVERSE EVENTS:
Time Frame: Baseline, 56 weeks
Description: The safety analysis set includes all randomized subjects who took study drug and were assessed by investigator after their first dose, whether or not they discontinue the study. Treatment-emergent adverse events were defined as events that started or worsened in the double-blind treatment phase after the first dose and before 7 days post last dose.
Arm/Group | NB16 | NB32 | Placebo
Serious Adverse Events (participants affected / at risk) | 9/569 | 9/573 | 8/569
Other Adverse Events (participants affected / at risk) | 345/569 | 365/573 | 230/569
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NB16 (N=569) | NB32 (N=573) | Placebo (N=569)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Hepatitis cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Whiplash injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cervical myelopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NB16 (N=569) | NB32 (N=573) | Placebo (N=569)
Constipation (Gastrointestinal disorders) | 90 (99) | 90 (98) | 32 (36)
Diarrhoea (Gastrointestinal disorders) | 31 (38) | 26 (28) | 28 (33)
Dry mouth (Gastrointestinal disorders) | 42 (44) | 43 (44) | 11 (12)
Nausea (Gastrointestinal disorders) | 155 (182) | 171 (197) | 30 (32)
Vomiting (Gastrointestinal disorders) | 36 (51) | 56 (63) | 14 (14)
Nasopharyngitis (Infections and infestations) | 32 (40) | 29 (33) | 31 (33)
Sinusitis (Infections and infestations) | 34 (39) | 30 (34) | 34 (39)
Upper respiratory tract infection (Infections and infestations) | 49 (62) | 57 (77) | 64 (83)
Dizziness (Nervous system disorders) | 44 (52) | 54 (65) | 15 (17)
Headache (Nervous system disorders) | 91 (107) | 79 (91) | 53 (58)
Insomnia (Psychiatric disorders) | 36 (38) | 43 (44) | 29 (30)
Hot flush (Vascular disorders) | 13 (15) | 30 (33) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If not already published by Sponsor as part of a multi-center publication, 18 months after conclusion of the study at all study centers, PI may publish the results for PI's study center individually. Prior to such publication, PI must provide Sponsor with at least 60 days to review and comment on the proposed publication. The review period may be extended by an additional 30 days upon request. Sponsor may delay publication for up to an additional 6 month period to file for patent protection.